CLINICAL TRIAL: NCT03678675
Title: Increased Ketorolac Administration After Cesarean Section and Its Effect on Opioid Use: a Randomized Control Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ketorolac Pain Study
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Results first posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-07

CONDITIONS: Post-operative Pain; Post-partum Pain; Cesarean Section Complications
Keywords: ketorolac; opiate; cesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The subjects, care providers, and investigators will be blinded to the assignments of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Protocol (No Intervention): Subjects randomized to the standard group will receive the standard postoperative pain protocol that is currently used at Tufts Medical Center. It includes two doses of IV Ketorolac every 6 hours as needed for postoperative pain. Ibuprofen would be ordered 6 hours following the last dose after the last study drug.
- Ketorolac Protocol (Experimental): Subjects randomized to the Ketorolac protocol will receive the study postoperative pain protocol. This includes 6 doses of IV Ketorolac, scheduled every 6 hours. The first dose is administered in the operating room or post-operative care unit.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — The intervention is a protocol of scheduled IV Ketorolac administered postoperatively.
  Arms: Ketorolac Protocol

SUMMARY:
To evaluate the efficacy of increased ketorolac in reducing opioid use after cesarean section.

DETAILED DESCRIPTION:
This was a single-center, randomized, double-blind, parallel-group trial to assess pain management following cesarean section with increased ketorolac versus placebo. All patients undergoing cesarean section with neuraxial anesthesia received two doses of 30mg IV ketorolac postoperatively per hospital protocol and were then randomized to receive an additional four doses of 30 mg of IV ketorolac or placebo every 6 hours. The primary outcome was the total morphine milligram equivalents (MME) used in the first 72 postoperative hours. Secondary outcomes included the number of patients that used no opioid postoperatively, postoperative pain scores, postoperative change in hematocrit and creatinine, and postoperative satisfaction with inpatient care and pain management. A sample size of 74 per group (n=148) was planned.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for care at Tufts Medical Center as an outpatient in obstetrics clinic or on Labor and Delivery.
* The subject must have had a cesarean section for any indication at Tufts Medical Center to be randomized to the study
* The subject is willing to have a phone call follow up conversation 2 weeks after their surgery.

Exclusion Criteria:

* Patients with allergy to ketorolac, NSAIDS or aspirin
* Patients with peptic ulcer disease, preexisting kidney or liver disease.
* Duramorph is not used as the anesthetic for the spinal/epidural during the cesarean section.
* Patient is hemodynamically unstable due to hemorrhage.
* Patient requires therapeutic anticoagulation in the post-operative period
* Patients with peripartum cardiomyopathy
* Provider decision to exclude patient.
* Patient diagnosis of chronic hypertension, gestational hypertension, preeclampsia, HELLP syndrome, or eclampsia
* A study subject may participate in another research study while participating in this research study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hostage J, Kolettis D, Sverdlov D, Ludgin J, Drzymalski D, Sweigart B, Mhatre M, House M. Increased Scheduled Intravenous Ketorolac After Cesarean Delivery and Its Effect on Opioid Use: A Randomized Controlled Trial. Obstet Gynecol. 2023 Apr 1;141(4):783-790. doi: 10.1097/AOG.0000000000005120. Epub 2023 Mar 9. PMID 36897140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Protocol | Ketorolac Protocol
Started | 74 | 74
Completed | 74 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Protocol | Ketorolac Protocol | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5) | 32.6 (5.2) | 32.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 4 | 6 | 10
  Race/Ethnicity: Black | 15 | 8 | 23
  Race/Ethnicity: Hispanic | 15 | 14 | 29
  Race/Ethnicity: White | 32 | 37 | 69
  Race/Ethnicity: Not reported | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 74 | 74 | 148

OUTCOME MEASURES:

1. Primary Outcome: The Total Morphine Milligram Equivalents (MME) Used in the First 72 Postoperative Hours
Description: The amount of MME's will be monitored for each group. MME's will be determined by the amount of opiate mediations administered. The MME value can range from 0 to typically 200 MME's, however there is no upper limit of measureable MME's. The MME's for each patient will be a sum of MME's administered throughout the course of the hospitalization.
Time Frame: Within 72 postoperative hours
Measure: Median (Inter-Quartile Range); unit: MME
Groups:
- Standard Protocol: Subjects randomized to the standard group will receive the standard postoperative pain protocol that is currently used at Tufts Medical Center. It includes two doses of IV Ketorolac every 6 hours as needed for postoperative pain.
- Ketorolac Protocol: Subjects randomized to the Ketorolac protocol will receive the study postoperative pain protocol. This includes 5 doses of IV Ketorolac, scheduled every 6 hours. The first dose is administered in the operating room.
  Ketorolac: The intervention is a protocol of scheduled IV Ketorolac administered postoperatively.
Arm/Group | Standard Protocol | Ketorolac Protocol
Number analyzed (Participants) | 74 | 74
MME | 60.0 [30 to 112.5] | 30 [0.0 to 67.5]

2. Secondary Outcome: Number of Participants With a Pain Score Greater Than 3
Description: The patient reported pain scores will be recorded and analyzed for each group. The Pain Score is determined by the patient using a visual analog scale with a range from 0-10, where 0 is no pain at all and 10 is the worst pain imaginable for the patient. Pain scores were collected by postpartum nursing staff per institutional policy. The number of patients with a pain score greater than 3 will be reported. A pain score greater than 3 was chosen as a cutoff as this is the pain score at which an opioid may be indicated for analgesia at our institution.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Protocol | Ketorolac Protocol
Number analyzed (Participants) | 74 | 74
Participants | 40 | 19

3. Secondary Outcome: The Number of Patients That Used no Opioid Postoperatively
Description: The number of patients in each arm that required no opioids for pain control postoperatively.
Time Frame: Within 72 post-operative hours
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Protocol | Ketorolac Protocol
Number analyzed (Participants) | 74 | 74
Participants | 24 | 9

4. Secondary Outcome: Postoperative Change in Hematocrit
Description: The change in patient hematocrit from baseline to POD1
Time Frame: Change in pre-operative hematocrit to POD1 hematocrit
Population: Post-operative day 1 hematocrit was available on 72 patients in the standard group and 73 patients in the ketorolac group.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | Standard Protocol | Ketorolac Protocol
Number analyzed (Participants) | 72 | 73
percentage of red blood cells in blood | -5.5 (3.5) | -5.5 (2.6)

5. Secondary Outcome: Change in Creatinine
Description: The change in patient's creatinine from POD1 to POD2
Time Frame: Change in creatinine from POD1 to POD2
Population: Post operative day 1 and 2 creatinine was collected on 68 patients in the standard group and 65 patients in the ketorolac group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard Protocol | Ketorolac Protocol
Number analyzed (Participants) | 68 | 65
mg/dL | .03 (.05) | .59 (.01)

6. Secondary Outcome: Postoperative Satisfaction With Inpatient Pain Control
Description: Two weeks after cesarean section, subjects were contacted by telephone to complete a survey on postpartum pain management. At least three attempts were made to contact subjects by telephone. In the follow-up phone call, patients were asked to rate their satisfaction with their postpartum care: very satisfied, satisfied, neutral, dissatisfied, or very dissatisfied. The number below describes the number of patients who reported they were "very satisfied" with their care.
Time Frame: Inpatient pain control satisfaction as reported at two weeks postpartum
Population: 52 patients in the standard protocol and 52 patients in the ketorolac group responded to the 2 week postpartum survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Protocol | Ketorolac Protocol
Number analyzed (Participants) | 52 | 52
Participants | 35 | 29

7. Secondary Outcome: Postoperative Satisfaction With Their Inpatient Postpartum Care.
Description: Two weeks after cesarean section, subjects were contacted by telephone to complete a survey on their overall postpartum care. At least three attempts were made to contact subjects by telephone. In the follow-up phone call, patients were asked to rate their satisfaction with their postpartum care: very satisfied, satisfied, neutral, dissatisfied, or very dissatisfied. The number below describes the number of patients that reported they were very satisfied with their care.
Time Frame: Satisfaction with inpatient care as reported at two weeks postpartum
Population: 52 patients in the standard protocol and 52 patients in the ketorolac group responded to the 2 week postpartum survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Protocol | Ketorolac Protocol
Number analyzed (Participants) | 52 | 52
Participants | 39 | 39

ADVERSE EVENTS:
Time Frame: Up to 6 weeks postpartum
Arm/Group | Standard Protocol | Ketorolac Protocol
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/74 | 1/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Protocol (N=74) | Ketorolac Protocol (N=74)
Headache (Nervous system disorders) | 0 (0) | 1 (1) — One patient in the ketorolac group was admitted postpartum with a headache.
Endometritis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — One patient in the placebo group developed endometritis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT03678675/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03678675/ICF_001.pdf